CLINICAL TRIAL: NCT01482858
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Analgesic Effects of the Gastrolith, in Osteoporotic Patients Suffering From Recent Skeletal Pain Caused by Vertebral Fractures
Brief Title: Analgesic Effects of the Gastrolith, in Osteoporotic Patients Suffering From Recent Skeletal Pain Caused by Vertebral Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMCS-003
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized double-blind multicenter study evaluating the safety of GASP and its analgesic effect on pain resulting from OCVF following oral administration of GASP vs. placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In this study the oral calcium treatments are blinded. The subjects, the investigators and any personnel involved in subjects' assessment, monitoring, analysis and data management will be blinded to the subject formulation assignment except the Sponsor who will be responsible for preparing, dispensing and labeling the investigational product IP. Blinded labels will be affixed to the vials prior to dosing by the un-blinded Sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrolith (Experimental): Gelatin capsules, each containing 500 mg of GASP (comprised of 125 ±5 mg elemental calcium) for oral use.
  Interventions: Dietary Supplement: Gastrolith
- Placebo (Placebo Comparator): Gelatin capsules, each containing 500 mg [comprised of 312.5 mg calcium carbonate (125 ±5 mg elemental calcium) and 187.5 mg of sucrose] for oral use as placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Gastrolith — Gelatin capsules, each containing 500 mg of GASP (comprised of 125 ±5 mg elemental calcium) for oral use.
  Arms: Gastrolith
Other: Placebo — Gelatin capsules, each containing 500 mg [comprised of 312.5 mg calcium carbonate (125 ±5 mg elemental calcium) and 187.5 mg of sucrose] for oral use as placebo
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety and analgesic effect (efficacy) of Gastrolith powder (GASP) on skeletal pain caused by osteoporotic vertebral compression fractures (OVCF) versus placebo, primarily as assessed by the Numeric Rating Scale (NRS), and Brief Pain Inventory (BPI). It is also intended to evaluate disability change with the Oswestry Low Back Pain Disability Index (ODI) and to evaluate whether GASP consumption leads to reduction in analgesic standard of care (ASOC) versus placebo, using weekly analgesic consumption diaries.

DETAILED DESCRIPTION:
Eighty (80) Osteoporotic subjects with recent reported severe back pain caused by OVCF will be blindly randomized into two groups (n=40 each). One group will receive GASP and the other Placebo.

The analgesic effect of GASP on top of the ASOC will be evaluated using weekly NRS and BPI assessments and three ODI questionnaires. Daily ASOC consumption will be monitored using weekly analgesic consumption diaries.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients aged 18-80 years old, inclusive.
* Diagnosed Osteoporotic vertebral compression fracture(s) in at least one vertebra caused by an atraumatic event or a minimal traumatic event such as falling from standing height or less, or by other minimal trauma besides a fall (see section 4.2 Table I for definitions), and visible by either X-ray radiography, CT or MRI.
* At least six (6) weeks and no more than six (6) months from the onset of severe back pain suspected to be caused by the OVCF.
* Presenting a score of ≥5 in the pain NRS during movement (getting up from a chair).
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Subject that had signed the ICF.

Exclusion Criteria:

* More than six (6) months from the onset of severe back pain suspected to be caused by OVCF.Subjects after vertebroplasty or kyphoplasty.
* Hypercalcemic subjects (calcium > 10.50 mg/dL).
* Subjects with renal diseases.
* Subjects with active malignancy or other active metabolic bone disease which is not osteoporosis.
* Subjects with cognitive impairments.
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Reduction of pain assessed by change in NRS from baseline to end of the trial | from baseline to end of the trial
  • Change from baseline to end-of-trial on NRS during movement (scale of 0 to 10) computed as follows.
  NRSchange = NRS42 - NRS0 NRS42 - NRS score at day 42 (end-of-trial) NRS0 - NRS score at day 0 (baseline)

SECONDARY OUTCOMES:
Reduction of pain assessed by change in BPI from baseline to end-of-trial | baseline to end-of-trial
  The BPI uses 0 to 10 numeric rating scales for item rating because of its simplicity, lack of ambiguity and seemed the best to use for cross-linguistic pain measurement. Since pain can be quite variable over a day, the BPI asks subjects to rate their pain at the time of responding to the questionnaire (pain now), and also at its worst, least, and average over the previous week. The ratings can also be made for the last 24 hours.
Reduction of disability assessed by change in ODI from baseline to end-of-trial | baseline to end-of-trial
  Oswestry Low Back Pain Disability Questionnaire - comprises of 10 sections describing the pain and its impact, each scored from 0 to 5 with higher values indicating more severe impact.
Reduction of ASOC assessed by weekly change in analgesic consumption diaries from baseline to end of trial | baseline to end of trial
  Analgesic drug consumption will be daily self-recorded by subjects in a diary bearing drug's name and daily dose. The number of tablets taken each day will be noted in each category.
All adverse events and serious adverse events will be collected and reported | Baseline until four (4) weeks after completion of the study.
  An adverse event is any untoward medical sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of the IPs whether or not considered as IP related. A new condition or the worsening of a pre-existing condition will be considered an AE. All abnormal findings considered to be clinically significant must be recorded as adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Eliad Davidson, MD, Principal Investigator — Hadassah Ein Carem Medical Center, Jerusalem, Israel
Locations (5):
- Israel (5):
  - Clalit Health Services - South District, Beersheba
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Ein Carem, Jerusalem
  - Sourasky Medical Center, Tel Aviv